CLINICAL TRIAL: NCT05404438
Title: Improvement of Mouth Breathing Habits During Sleep in Patients With Obstructive Sleep Apnea
Brief Title: Mouth Breathing Habits Improvement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: YM107083E
Record Dates: First submitted 2022-05-16; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2018-09

CONDITIONS: OSA
Keywords: mouth breathing; mouth puffing; sleep apnea; oral appliance
MeSH Terms: conditions — Mouth Breathing; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): single arm study
  Interventions: Other: Oral Appliances

INTERVENTIONS:
Other: Oral Appliances — A pre-experimental, single-group pretest-posttest design was performed. At stage one, each participant underwent a 2-day general sleeping test and a 2-day sleeping test with mouth tape. At stage two, participants underwent conventional impressions for TPD and TED appliances and were then randomly assigned to wear the TPD or TED; together for two days of sleeping test with their mouth taped. After a 2-day break (washout), with the same procedure, participants wore the other appliance for another 2-day sleeping test and decided accordingly the optimal appliance that had reduced their ODI scores more. At stage three, participants wore their optimal appliance mouth-taped during sleep for 6 weeks. At the end of the intervention, all participants underwent few days sleeping test for final results.

SUMMARY:
This study intends to investigate the improvement in patients with OSA through objective measurement, including oxygen desaturation index (ODI) and the percentage reduction in intermittent mouth puffing (IMP) before and after the intervention. The oral appliances are placed between the tongue and the soft palate to reduce the oral ventilation space. A total of 24 participants aged between 36 and 57 years were identified with ODI above 5 events/hour by measuring their blood oxygen and with an originally designed mouth puffing detector to find out those who were still mouth-puffed when their mouths were taped. A suitable appliance was chosen for the participants between the two originally designed oral appliances, tongue pressed device (TPD) and tongue elevated device (TED), and the intervention lasted for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 20-60 years old,
* (2) having symptoms of OSA including snoring, daytime sleepiness, etc.
* (3) AHI & ODI >=5 events/hour,

Exclusion Criteria:

* (1) taken sleep medication within the last two months or were on long-term use,
* (2) reported tobacco, alcohol, caffeine or drug addiction,
* (3) cancer, cardiovascular disease, psychiatric illness, kidney disease, diabetes mellitus, or other sleep disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Differences in OSA-related variables before and after the six weeks oral device intervention | baseline, six weeks after intervention
  According to OSA-related variables, we can analyze participants' ODI (events/hours), mean SpO2 (%), the lowest SpO2(%), and the percentage of total record time with oxygen saturation below 90% (T90) to evaluate their objective sleep quality.
Differences in percentage of mouth puffing before and after the six weeks oral device intervention | baseline, six weeks after intervention
  According to the number of mouth puffing by minutes, mouth puffing signals were divided into four types, including non-mouth puffing (NMP, no or less than 3 times MPSs on both sides), complete mouth puffing (CMP, regularly MPS on both sides, usually above 8-10 times), intermittent mouth puffing (IMP, irregularly MPS in both side, usually between 3-8 times), and side mouth puffing (SMP, showing one-side MPSs) to evaluate the percentage of mouth breathing while sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl CH Yang, professor, Study Chair — Institute of Brain Science ,National Yang-Ming University, Taipei City, Taiwan
Locations (1):
- Faculty of Medicine, and Institute of Brain Science, National Yang-Ming Chiao-Tung University, Taipei, Taiwan